CLINICAL TRIAL: NCT02192879
Title: A Comparison of the Efficacy of Alternative Analgesia Modalities in Complex Hepatic Resection Surgery: Thoracic Epidural Analgesia Versus Continuous Paravertebral Block With Patient-Controlled Analgesia Versus Patient-Controlled Analgesia
Brief Title: TEA vs. PVB vs. PCA in Liver Resection Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042166
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Pain Management Strategies in Liver Resection Surgery
Keywords: thoracic epidural; continuous paravertebral catheter; PCA; liver resection; pain management
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thoracic Epidural (Active Comparator)
  Interventions: Device: thoracic epidural
- Continuous Paravertebral Catheter (Active Comparator)
  Interventions: Device: continuous paravertebral catheter
- Patient-Controlled Analgesia (Active Comparator)
  Interventions: Drug: Patient-Controlled Analgesia

INTERVENTIONS:
Device: thoracic epidural — Thoracic Epidural catheters will be placed between T8-12 interspaces preoperatively. Epidural hydromorphone (200-600mcg) will be given preoperatively. TEA will be dosed intraoperatively with a continuous infusion of 0.25% bupivacaine at 3-6ml per hour. At the end of surgery, infusion will be changed to 0.125% bupivacaine + 10mcg/ml hydromorphone at 4-6ml/hour. In PACU, a PCEA button will given to the patient for bolus dosing of 1-2ml and a lockout of 30 minutes. Changes to the epidural infusion solution, rate, and PCEA bolus dosing will be made clinically as required by the Acute Pain Service (APS).
  Arms: Thoracic Epidural
Device: continuous paravertebral catheter — Bilateral PVB catheters will be placed between the T8-12 interspaces preoperatively. 10ml of 0.5% ropivacaine will be injected into the paravertebral space, then catheter placed. The same procedure will be used for the placement of the PVB catheter on the opposite side. The catheter may be bolused with 5ml 0.5% ropivacaine hourly intraoperatively if needed. In PACU, PVB catheters will be infused continuously with 0.2% ropivacaine at 8-12ml/hr. Subjects will also be given a hydromorphone PCA button to deliver additional IV opioid medication to the patient as needed.
  Arms: Continuous Paravertebral Catheter
Drug: Patient-Controlled Analgesia — Intravenous hydromorphone PCA will be initiated postoperatively with dosing prescriptions made by the primary surgical team.
  Arms: Patient-Controlled Analgesia

SUMMARY:
This study aims to compare the efficacy and safety of three alternative methods of analgesia in patients undergoing complex liver resection surgery: 1) thoracic epidural analgesia (TEA), 2) continuous paravertebral block (PVB) with patient-controlled analgesia (PCA) and 3) patient-controlled analgesia (PCA) alone. Regional anesthesia techniques such as TEA and PVB may improve recovery and decrease postoperative pain scores in addition to other benefits such earlier return of bowel function and shortened length of hospital stay, although some practitioners have voiced concerns about the safety and efficacy of these techniques in patients after liver resection who may develop postoperative coagulation abnormalities. The investigators plan to enroll a total of 150 patients (adults >/= 18 years of age who meet study criteria) scheduled for complex liver resection surgery in this study, who will then be randomized into 50 patients per arm of the study (3 total arms). Postoperative pain scores will be collected in PACU and throughout the patient's hospital stay as well as routine blood tests including complete blood count, coagulation labs (PT/INR, aPTT) and serum creatinine to measure renal function. The study team will also collect additional data prospectively on all patients enrolled in the study; these parameters will include age, sex, type of operation performed, length of operation, volume of intraoperative blood loss, volume of intraoperative fluid administration including blood products, daily postoperative intravenous fluid administration, length of time to first feeding, day of epidural catheter removal, length of hospital stay and incidence of major postoperative complications (surgical, respiratory, cardiac, renal, etc.). Once primary and secondary data points are obtained, the data will undergo rigorous statistical analysis using the appropriate statistical techniques to determine the outcomes. The investigators propose that epidural and/or paravertebral analgesia may improve recovery times and decrease hospital length of stay, which would be beneficial for the patient as well as decrease hospital costs. In addition, if better postoperative pain management scores can be achieved with epidural or paravertebral analgesia, and no significant prolonged postoperative coagulopathy is associated with patients undergoing major hepatic resection surgical procedures, these regional analgesia strategies can be considered a safe option for pain management in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years and </= 80 years
* Scheduled for elective hepatic resection surgery

Exclusion Criteria:

* Preexisting coagulopathy (INR >1.5)
* Spinal stenosis
* Local infection in area where catheter will be inserted
* Severe cardiovascular disease (NYHA Class III/IV)
* Severe pulmonary disease (FEV1 <50% of predicted value)
* Allergy or sensitivity to narcotics or local anesthetics
* BMI >45
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Malinzak, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Started | 3 | 4 | 3
Completed | 3 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia | Total
Number analyzed (Participants) | 3 | 4 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 9
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Highest VAS Pain Score at Rest
Description: Post-operative pain scores at rest, as assessed by Pain Assessment Scales (Wong-Baker Faces Scale and Visual Analog Pain Scale (VAS) will be the primary outcome measured. Pain scores will be collected per standard PACU protocol (every 60 minutes) and on the hospital ward at hours 2, 4, 6 and 12, and then daily until day 3 or when the epidural/paravertebral catheter is removed. Postoperative pain at rest will be defined as the highest VAS pain score reported by each patient at any time. Pain score is from 0 (no hurt) to 10 (hurts worst).
Time Frame: postoperatively until regional catheter removed, with an expected average of 3 days and up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
units on a scale | 5.67 (2.08) | 7.0 (2.94) | 7.67 (2.51)

2. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay will be recorded for each of the 3 groups to see if there is a statistical difference between groups.
Time Frame: time to discharge after surgery, with an expected average of approximately 7-10 days, up to 6 weeks if complications arise
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
days | 10.33 (4.93) | 6.25 (2.5) | 7.0 (1.0)

3. Secondary Outcome: Gastrointestinal Recovery
Description: Postoperative return of bowel function and time to first feeding will be recorded for each of the 3 groups.
Time Frame: postoperatively until return of bowel function, up to 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
days | 4.33 (0.58) | 4.25 (2.63) | 5.33 (1.53)

4. Secondary Outcome: Cumulative Postoperative Opioid Requirement
Description: Cumulative postoperative opioid use in morphine equivalents will be recorded for subjects in the 3 arms of the study. The investigators hypothesize that the TEA and/or PVB arms may show less opioid use over PCA.
Time Frame: postpoperatively until regional catheter removed or subjects transitioned to an oral pain management regimen, an expected average of 3 days and up to 7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
mg | 388.33 (430.71) | 224.6 (236.5) | 176.20 (40.14)

5. Secondary Outcome: Incidence of Major Postoperative Complication
Description: Major surgical, infectious, respiratory, cardiac, and renal complications will be recorded for subjects in each arm of the study.
Time Frame: as for outcome 2
Measure: Number; unit: complications
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
complications | 2 | 2 | 0

6. Secondary Outcome: Highest VAS Pain Scores With Coughing
Description: Post-operative pain scores with coughing, as assessed by Pain Assessment Scales (Wong-Baker Faces Scale and Visual Analog Pain Scale (VAS) will be measured. Pain score is from 0 (no hurt) to 10 (hurts worst).
Time Frame: postoperatively until regional catheter removed, with an expected average of 3 days and up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 3
units on a scale | 7.33 (2.52) | 8.0 (2.45) | 8.33 (1.53)

7. Other Pre Specified Outcome: Serious Adverse Events Associated With Regional Catheter Placement
Description: Serious adverse events in the 2 arms with regional catheters (TEA and PVB) will be monitored
Time Frame: postoperatively until removal of regional catheter removed, with an average of 3 days up to 7 days
Population: only patients who had a catheter
Measure: Number; unit: serious adverse events
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Number analyzed (Participants) | 3 | 4 | 0
serious adverse events | 0 | 0 |

ADVERSE EVENTS:
Arm/Group | Thoracic Epidural | Continuous Paravertebral Catheter | Patient-Controlled Analgesia
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thoracic Epidural (N=3) | Continuous Paravertebral Catheter (N=4) | Patient-Controlled Analgesia (N=3)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
diaphragm leak (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
bile leak (Gastrointestinal disorders) | 1 | 0 | 0
blurred vision (Eye disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Unable to recruit adequate number of participants, and decision was made to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes